CLINICAL TRIAL: NCT02793999
Title: Perinatal Brain Injury: Potential of Innovative NIRS to Optimize Hypothermia
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ellen Grant, Professor of Radiology, Boston Children's Hospital
Other Study IDs: P00012473; R01HD076258-02 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-06-08 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypoxic Ischemic Brain Injury; Neonatal Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Near-Infrared Spectroscopy (NIRS)

SUMMARY:
The purpose of this study is to improve the ability of the investigators to monitor brain health in newborn babies at risk of brain injuries. The researchers will be using an investigational system of devices to non-invasively (that, is, without penetrating the skin), measure the amount of oxygen going to and being used by the brain. They will be taking some bedside research measurements during the babies' stay at the hospital. With these measurements, the intention is to study the role of oxygen in brain injury and test the efficacy of the research device and its potential as a permanent bedside diagnostic device.

DETAILED DESCRIPTION:
Neonatal encephalopathy (NE) due to hypoxia-ischemia is a major public health concern as it occurs in 6/1000 live term births and has devastating consequences. Many affected neonates suffer lifelong motor disabilities and epilepsy, but increasingly the high prevalence of cognitive and behavioral disabilities is becoming appreciated. In hypoxia-ischemia there is a decrease in blood and oxygen delivery, followed by reperfusion with transient energy recovery. What follows is a "window of opportunity" where excitotoxicity and associated increased cerebral metabolism eventually lead to secondary energy failure and irreversible cell death. In this window, therapeutic hypothermia (TH) is currently the only treatment available with proven efficacy. TH acts primarily by decreasing cerebral metabolism, thus preserving energy stores.

Although the current gold standard for brain injury detection is magnetic resonance imaging (MRI), MRI is impractical as a screening tool and cannot provide bedside monitoring to optimize individual responses to therapies. Commercially available continuous wave (CW) near infrared spectroscopy (NIRS) systems provide bedside measures of cerebral oxygen saturation (SO2) but SO2 alone cannot assess oxygen metabolism, as oxygen delivery is not taken into account. What is needed is a bedside tool that can monitor cerebral metabolism to detect elevations in metabolism that suggest evolving hypoxic-ischemic injury, and decreases in metabolism that suggest response to therapy. Cerebral oxygen consumption (CMRO2) is a direct measure of cerebral metabolism and therefore the investigators propose to measure an index of CMRO2 at the bedside using the innovative combination of Frequency Domain Near-Infrared Spectroscopy (FDNIRS) and Diffuse Correlation Spectroscopy (DCS). The initial studies from the investigators show that CMRO2 is elevated in neonates with MRI evidence of perinatal brain injury, and confirm that neonates on TH have significantly lower CMRO2 than normal controls. Following these exciting results, they now propose a feasibility study to determine if FDNIRS-DCS can screen for involvement, assess response to treatment, and predict outcomes in one of the largest neonatal populations requiring early screening and immediate intervention: neonatal encephalopathy. To assess early outcomes, the research team proposes an innovative combination of advanced neurobehavioral testing, regional FDNIRS-DCS measures and quantitative MRI analysis using MRIs obtained without sedation. If the hypotheses prove true, it will help in determining if bedside indices of CMRO2 provided by FDNIRS-DCS can optimize TH for individual neonates, thereby improving neurodevelopmental outcomes. Success at this stage will also allow exploration of the potential for FDNIRS-DCS to determine the additional benefits of emerging new treatments for NE and to screen for other treatable neonatal disorders.

ELIGIBILITY:
Inclusion criteria:

Neonates must be > 33 weeks gestational age (GA) and meet inclusion criteria for one of the two groups:

1. Therapeutic Hypothermia (TH) Group:

   1. Undergo TH as part of their clinical management
   2. Parents consent to multiple measures in the first week of life.
2. No Therapeutic Hypothermia (no-TH) Group:

   1. Signs will be defined broadly as any one of the following which can be considered evidence of NE caused by HIE or other etiologies: i) Seizures alone or ii) any of the following: abnormal consciousness, difficulty maintaining respiration, difficulty feeding (presumed central origin), abnormal tone or reflexes.
   2. Parents consent to multiple measures in the first week of life.

Exclusion criteria:

Exclusion criteria includes neonates born at GA ≤ 33 weeks or < 2.0 kg, with implanted devices or other devices that preclude the use of MRI will be excluded from the follow up MRI session.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates must be > 33 weeks gestational age (GA) and meet inclusion criteria for one of the two groups:
  1. Therapeutic Hypothermia (TH) Group:
     1. Undergo TH as part of their clinical management
     2. Parents consent to multiple measures in the first week of life.
  2. No Therapeutic Hypothermia (no-TH) Group:
     1. Signs will be defined broadly as any one of the following which can be considered evidence of NE caused by HIE or other etiologies: i) Seizures alone or ii) any of the following: abnormal consciousness, difficulty maintaining respiration, difficulty feeding (presumed central origin), abnormal tone or reflexes.
     2. Parents consent to multiple measures in the first week of life.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2015-05; Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Compare metrics such as hemoglobin oxygen saturation and cerebral metabolic rate of oxygen consumption as obtained from novel NIRS technology in neonates at risk for brain injury to normal controls. | early inpatient phase (0-2 months of age)
  The infants undergoing treatment with therapeutic hypothermia (TH) and those who are identified with neonatal brain injury but are not candidates for TH will be compared. Both groups will also be compared to normal controls.

SECONDARY OUTCOMES:
Perform NIRS, MRI and Neurodevelopmental testing (using Bayley Scales for Infant Development) between 2-12 months. | up to 12 months of age
  Explore correlations between all NIRS and MRI measures, and neurodevelopmental outcome at 2-12 months.
Perform Neurodevelopmental testing at 16-24 months using Bayley Scales for Infant Development. | up to 24 months of age
  Explore correlations between all NIRS and MRI measures, and neurodevelopmental outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ellen Grant, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No